CLINICAL TRIAL: NCT01043341
Title: Knowledge and Attitude About HPV Vaccines Among Women
Brief Title: Knowledge and Attitude About HPV Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Sylvia Michelina Fernandes Brenna, Universidade Cidade de São Paulo
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: HPV vaccines
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Knowledge; Attitude; Behavior
Keywords: HPV; vaccines; knowledge; attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- behavioral (Active Comparator): the women received a folder about HPV infection and vaccines and answered a questionaire about sexual behavior, HPV infection and vaccines.
  Interventions: Behavioral: educative folder
- no intervention (No Intervention): the women answered a questionaire about sexual behavior, HPV infection and vaccines
  Interventions: Behavioral: educative folder

INTERVENTIONS:
Behavioral: educative folder — folder about HPV infection and vaccines
  Other Names: HPV vaccines information

SUMMARY:
The purpose of this study was to analyze the knowledge and attitude about HPV vaccines among Brazilian women after an educative intervention. The knowledge was measured on sexual behavior and HPV infection. The attitude was measured on acceptance of vaccines.

DETAILED DESCRIPTION:
Two hundred Brazilian women were selected ranged 18 to 30 years old. They were randomized on two groups: 1) One hundred received a brief educative intervention about HPV infection and vaccines and answered a questionaire about sexual behavior, HPV infection and vaccines and 2)one hundred not received anything and answered the same questionaire.

ELIGIBILITY:
Inclusion Criteria:

* healthy women

Exclusion Criteria:

* previous CIN or cervical cancer treatment

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Incorrect knowledge about HPV vaccines was detected on more than 50% women, however the attitude to accept the HPV vaccine was improved after educative intervention. | 2 years

SECONDARY OUTCOMES:
The acceptance of HPV vaccines by the women was depended on the sponsor by the public heath services | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia MF Brenna, MD, PHD, Study Director — Universidade Cidade de São Paulo; Kari J Sirjanen, MD, PhD, Study Chair — University of Turku
Locations (1):
- Universidade Cidade de São Paulo, São Paulo, São Paulo, Brazil